CLINICAL TRIAL: NCT03406806
Title: Comparison of the Gaitbox, SprintSystem Device and NIH Toolbox 4 Meter Walk
Brief Title: Gaitbox Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00089655
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-03

CONDITIONS: Validation of Gait Speed Device Against Existing Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GaitBox (Experimental)
  Interventions: Other: Gaitbox
- Sprint System device (Active Comparator)
  Interventions: Other: SprintSystem device
- NIH Toolbox 4 meter test (Active Comparator)
  Interventions: Other: NIH toolbox 4 meter walk

INTERVENTIONS:
Other: Gaitbox — The walking path will be set according to the directions of the NIH toolbox 4 meter clinic walk test which includes marking the beginning and end of the walking path. A standard manual stopwatch will be used to record time. The examiner will demonstrate the task then instruct the participant to "Walk at a comfortable pace" and count down by saying: "3, 2, 1, go." The stop watch will be used to time the amount of time it takes to walk between the cones. Subjects will complete 3 timed trials. The time will be recorded in the log. Simultaneously, the Sprint System [6] will be operated according to manufacturers instructions. The Gaitbox will be set up at the end of the 4 meter walking path at a height of 4 feet from the floor. Times/speeds will be recorded on log sheet.
  Arms: GaitBox
Other: SprintSystem device — The walking path will be set according to the directions of the NIH toolbox 4 meter clinic walk test which includes marking the beginning and end of the walking path. A standard manual stopwatch will be used to record time. The examiner will demonstrate the task then instruct the participant to "Walk at a comfortable pace" and count down by saying: "3, 2, 1, go." The stop watch will be used to time the amount of time it takes to walk between the cones. Subjects will complete 3 timed trials. The time will be recorded in the log. Simultaneously, the Sprint System [6] will be operated according to manufacturers instructions. The Gaitbox will be set up at the end of the 4 meter walking path at a height of 4 feet from the floor. Times/speeds will be recorded on log sheet.
  Arms: Sprint System device
Other: NIH toolbox 4 meter walk — The walking path will be set according to the directions of the NIH toolbox 4 meter clinic walk test which includes marking the beginning and end of the walking path. A standard manual stopwatch will be used to record time. The examiner will demonstrate the task then instruct the participant to "Walk at a comfortable pace" and count down by saying: "3, 2, 1, go." The stop watch will be used to time the amount of time it takes to walk between the cones. Subjects will complete 3 timed trials. The time will be recorded in the log. Simultaneously, the Sprint System [6] will be operated according to manufacturers instructions. The Gaitbox will be set up at the end of the 4 meter walking path at a height of 4 feet from the floor. Times/speeds will be recorded on log sheet.
  Arms: NIH Toolbox 4 meter test

SUMMARY:
The purpose of this study is to validate the walking velocity measured by the Gaitbox as compared to the measures obtained by clinicians administering the timed 4 meter walk test and the Sprint System device. The investigators have developed a compact device, the Gaitbox, which measures walking speed automatically. The device has an infrared light sensor that is capable to accurate distance measurements. To take a speed measurement, the device is placed at the end of the walking path and the subject simply walks towards the device. The device automatically records a starting and ending distance and calculates and displays walking speed in m/sec. This is a prospective, single site study. Up to 60 subjects will be enrolled at Duke. Subjects will be asked to complete the 4-meter walk test, three (3) times. Three speed measuring methods will be conducted simultaneously: NIH toolbox 4 meter clinic walk test and the Sprint System device (commercially available device typically used for timing track and field events), and the Gaitbox. The purpose is to validate the Gaitbox to the clinical NIH toolbox 4 meter test and against the Sprint System device. The following comparisons of speed will be made: Human timer 1 to human timer 2, Average human timer to Gaitbox, Gaitbox to Sprint System.

DETAILED DESCRIPTION:
This is a prospective, single site study. Up to 60 subjects will be enrolled at Duke. Subjects will be asked to complete the 4-meter walk test, three (3) times. Three speed measuring methods will be conducted simultaneously: NIH toolbox 4 meter clinic walk test and the Sprint System device (commercially available device typically used for timing track and field events), and the Gaitbox.

NIH toolbox 4 meter clinic walk test: The walking path will be set according to the directions of the NIH toolbox 4 meter clinic walk test which includes marking the beginning and end of the walking path. Tape will be used to mark beginning and end of timing section of the walking path to allow for acceleration and deceleration. A standard manual stopwatch will be used to record time. The examiner will demonstrate the task then instruct the participant to "Walk at a comfortable pace" and count down by saying: "3, 2, 1, go." The stop watch will be used to time the amount of time it takes to walk between the cones. Subjects will complete 3 timed trials. The time will be recorded in the log.

Simultaneously, the Sprint System will be operated according to manufacturers instructions. The device will be setup on tripods 4 feet from the floor so as to be triggered by the subject's torso rather than feet and set to measure data at the same distances as the gait box. The device will be set up to record times at the same distances as the Gaitbox. The Sprint System is used to time track running events by breaking two invisible light beams. Timing starts when the subject crosses the first line and stops when the second line is crossed. The times are displayed on a handheld display. Times will be transferred to the log sheet.

The Gaitbox will be set up at the end of the 4 meter walking path at a height of 4 feet from the floor. To operate, investigator presses reset button, waits for ready light and tells subject to go. Speed is measured automatically and result is displayed. Times/speeds will be recorded on log sheet.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 55 or older
* Subjects must be able to complete three 5 meter walks, with or without assistive device such as canes, crutches or walkers.

Exclusion Criteria:

* Subjects with a physical, cognitive, or behavioral impairment that would prevent the safe completion of the testing, or affect the ability to follow study directions will be excluded from participation.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Time of 4 meter walk test | Up to 1 hour
Speed of 4 meter walk test | Up to 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Caves, ME, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Background] Lusardi, Michelle M. (2012). "Is Walking Speed a Vital Sign? Absolutely." Topics in geriatric rehabilitation 28(2): 67-76.
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966
- [Background] Hardy SE, Perera S, Roumani YF, Chandler JM, Studenski SA. Improvement in usual gait speed predicts better survival in older adults. J Am Geriatr Soc. 2007 Nov;55(11):1727-34. doi: 10.1111/j.1532-5415.2007.01413.x. Epub 2007 Oct 3. PMID 17916121
- See also: NIH Toolbox: Assessment of Neurological and Behavioral Function — http://www.nihtoolbox.org
- See also: Sprint system — http://browertiming.com/products/tc-timing-system/